CLINICAL TRIAL: NCT07034911
Title: Impact of Sub-anaesthetic Dose of Ketamine Versus Ephedrine on Post Spinal Hypotension in Caesarean Delivery
Brief Title: Ketamine vs Ephedrine on Post Spinal Hypotension in Caesarean Delivery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FMASU MS130/2024
Record Dates: First submitted 2025-06-15; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2024-03

CONDITIONS: Post Spinal Hypotension
MeSH Terms: interventions — Ketamine; Ephedrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine group (Active Comparator): 0.5mg/kg ketamine
  Interventions: Drug: Ketalar
- Ephedrine group (Active Comparator): 15 mg ephedrine
  Interventions: Drug: Ephedrine

INTERVENTIONS:
Drug: Ketalar — women receiving sub-anesthetic dose of ketamine of 0.5 mg/kg IV bolus in 3 ml of normal saline.
  Other Names: Ketamine
  Arms: Ketamine group
Drug: Ephedrine — women receiving bolus of 15mg of ephedrine
  Arms: Ephedrine group

SUMMARY:
Comparing ketamine and ephedrine to decrease the incidence of post spinal hypotension after caesarean section delivery.

DETAILED DESCRIPTION:
To compare the effect of ketamine versus ephedrine in decreasing the incidence of hypotension in caesarean section delivery a study group including 50 participants will receive ketamine and 50 group will receive ephedrine after the consent and detailed history the two groups will receive preload of 500ml enter acetate then dormicum for sedation then spinal anesthesia will be performed initial blood pressure and heart rate will be measured then every five minutes

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Caesarian Section under spinal anesthesia,
* Patients aged 18-45 years,
* At term (≥37-week gestation),
* American Society of Anaesthesiologists (ASA) physical status 1 or 2 Exclusion Criteria:
* Pre-eclampsia,
* Chronic hypertension, cardiovascular troubles,
* Any contraindication to regional anesthesia such as local infection or bleeding disorders,
* Any hypersensitivity to ketamine.
* Declined informed consent.
* American Society of Anaesthesiologists (ASA) physical status lll or lV

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Incidence of hypotension post spinal in CS | From injection till the end of surgery
  For ketamine Group: women receiving sub-anesthetic dose of ketamine of 0.5 mg/kg IV bolus in 3 ml of normal saline. ( Reves JG et al,2010 )
  * For ephedrine Group: women receiving bolus of 15mg of ephedrine
  * All the patients will receive 2 mg midazolam IV directly after delivery of the fetus.( Perumal DK et al )
  * Heart Rate (HR) and Mean Arterial Blood Pressure (MAP) will be recorded at baseline 5 minutes prior to the intrathecal injection and 5 minutes, 10 minutes, 15 minutes, and 20 minutes after the injection and then every 15 minutes till the end of the operation.
  * Incidence of hypotension will be recorded which is defined as MAP less than 20% below the baseline or was ≤ 65 mmHg. Incidence of severe hypotension ≤ 50 mmHg will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Basant E Mohamed, M.B.B.CH, Principal Investigator — Anesthesia resident Alain Shams University
Locations (1):
- Ainshams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Before1/2026
Access Criteria: Free